CLINICAL TRIAL: NCT06841510
Title: A Prospective, Multicenter, Observational Study to Evaluate the Efficacy and Safety of GENOSS SES in Patients With Coronary Artery Disease
Brief Title: Efficacy and Safety of GENOSS SES in Patients With Coronary Artery Disease
Acronym: GENOSS SES
Status: Active, not recruiting | Type: Observational
Sponsor: Genoss Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-DS0501-09
Record Dates: First submitted 2025-02-17; First posted 2025-02-24 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-02

CONDITIONS: Coronary Arterial Disease (CAD)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GENOSS Sirolimus Eluting Coronary Stent System: patients with coronary artery disease treated with GENOSS SES

SUMMARY:
Efficacy and Safety of GENOSS SES in patients with coronary artery disease

DETAILED DESCRIPTION:
GENOSS SES

ELIGIBILITY:
Inclusion Criteria:

1. Patients of 19 and over
2. Patients with coronary artery disease treated with GENOSS SES
3. Participants who voluntarily decide to participate in this clinical trial, agree to the study protocol and clinical follow-up plan, and provide written informed consent as study participants

Exclusion Criteria:

1. Patients who are contraindicated in the use of heparin, aspirin, clopidogrel, sirolimus, cobalt chromium and contrast agents
2. Patients who are pregnant or planning to become pregnant
3. Patients with a planned surgery to discontinue antiplatelet agents within 12 months
4. Patients with a life expectancy of less than 1 year
5. Patient with cardiogenic shock at the time of hospitalization and had a low chance of survival based on medical judgment.
6. Patients who have already received treatment with another DES (Drug Eluting Stent) or BMS (Bare Metal Stent) at the time of registration
7. Patients participating in randomized controlled trials using other medical devices

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease treated with GENOSS SES
Sampling Method: Non-Probability Sample
Enrollment: 1118 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Device-oriented composite endpoint | at 12 months after the procedure
  DOCE is defined as a composite of cardiac death, target vessel-related myocardial infarction (TV-MI) and clinically indicated target-lesion revascularization (TLR).

SECONDARY OUTCOMES:
Patient-oriented composite endpoint | at 12 months after the procedure
  POCE is defined as a composite of all-cause death, any myocardial infarction, and any revascularization.
All-cause deaths | at 12 months after the procedure
Cardiac death | at 12 months after the procedure
Non-cardiac death | at 12 months after the procedure
Any myocardial infarction | at 12 months after the procedure
Target vessel-related myocardial infarction (TV-MI) | at 12 months after the procedure
Any revascularization | at 12 months after the procedure
Clinically indicated target lesion revascularization (TLR) | at 12 months after the procedure
Stent thrombosis | at 12 months after the procedure
Lesion success | during the procedure
  When the final residual lesion stenosis is less than 50% using any surgical method.
Procedure success | immediately after the procedure
  When the final residual lesion stenosis is less than 50% using any surgical method, and there is no post-procedure death, myocardial infarction, or revascularization during the hospitalization period.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No